CLINICAL TRIAL: NCT05508126
Title: Diagnostic Accuracy of Multi-parametric MRI and Dual-energy CT in Gastric Cancer: a Paired Validating Confirmatory Study
Brief Title: Multi-parametric MRI and Dual-energy CT in Patients of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-SR-475
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer Stage
Keywords: Computed Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary staging group I: All patients will be treated according to standard practice. Patients in group I are patients that will be stratified for radical gastrectomy or endoscopic resection. Group I will undergo only a primary staging. All patients will take DECT and mpMRI examination within 1 week before surgery.
  Interventions: Diagnostic Test: DECT examination; Diagnostic Test: mpMRI examination
- Restaging group II: Patients in group II are patients that will be stratified for neoadjuvant chemotherapy.
  Group II will undergo a primary staging (DECT and mpMRI) and 1-2 times restaging (DECT and mpMRI).
  Interventions: Diagnostic Test: DECT examination; Diagnostic Test: mpMRI examination

INTERVENTIONS:
Diagnostic Test: DECT examination — DECT examinations will be performed using a 192-slice CT scanner (SOMATOM, Force, Siemens, Forchheim, Germany).
Diagnostic Test: mpMRI examination — The examinations were conducted on a 3-T MR scanner (MAGNETOM Skyra; Siemens Healthcare, Erlangen, Germany).

SUMMARY:
Accurate preoperative staging of gastric cancer is of major importance for guiding therapeutic decision-making, preventing both under- and over-treatment. The purpose of this study is to investigate the diagnostic performance of the Multi-parametric magnetic resonance imaging (mpMRI) and dual-energy computed tomography (DECT) in gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is the leading cause of cancer-related death worldwide. The therapeutic approach to gastric cancer is strongly dependent on preoperative stage. The crucial role of gastric cancer imaging lies in implementing individualized treatment regimens according to various stages of tumor.

CT scanning has been recommended as the first-line image modality for preoperative evaluation of gastric cancer by the 8th AJCC staging manual. However, for traditional CT, the accuracy of staging is highly variable and the sensitivity of early gastric cancer detection is relatively low. Recently, DECT has been increasingly used in clinical practice due to its powerful post-processing technique. A recent small sample study showed that monoenergetic images at 40 KeV improved lesion depiction and higher T stage accuracy for gastric cancer. Therefore, this study chose DECT instead of traditional CT to explore the diagnostic performance in preoperative staging.

Historically, the role of MRI in gastric cancer has been limited, and the guidelines have not yet recommended MRI as a first-line examination scheme. But with the continuous technical improvements for abdominal imaging (e.g. breath-hold sequences and high Resolution diffusion-weighted imaging (DWI), free-breathing dynamic contrast-enhanced (DCE) sequence), mpMRI has become a promising imaging technology. In addition, given the advantages of non-radiation, non-invasiveness, and excellent soft tissue contrast, mpMRI may be more suitable for neoadjuvant therapy patients who require multiple evaluations.

Patients with gastric cancer confirmed by endoscopic biopsy will be prospectively included in this study. Patients undergo both mpMRI and DECT at baseline to stage the primary tumor, regional lymph nodes, and to rule out distant sites of disease. The interval between mpMRI and DECT examinations should not exceed 7 days. All patients will be treated according to standard practice in our institution. Patients receiving neoadjuvant chemotherapy will undergo mpMRI and DECT scan again for restaging. The postoperative pathology results of these two examination methods were prospectively collected, and their efficacy was calculated according to the reference standard. After completion of study intervention, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with preoperative pathologically confirmed GC by endoscopy and preoperative imaging data (DECT/mpMRI) were included.
* No contraindications for CT/MRI examination
* Written informed consent

Exclusion Criteria:

* Patients with a history of previous therapy.
* Patients with recurrent gastric cancer
* Patients with a history of severe allergy to contrast agents
* Patients with imaging artefacts affect the evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with gastric cancer by endoscopically biopsy will be considered for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DECT and mpMRI in tumor staging assessment | 2 years
  Accuracy for both imaging techniques in the prediction of tumor staging.
Diagnostic performance of DECT and mpMRI in tumor restaging assessment | 2 years
  Accuracy for both imaging techniques in the prediction of tumor restaging.

SECONDARY OUTCOMES:
The kappa value | 2 years
  Inter-rater reliability of the DECT and mpMRI in tumor assessment
Predictive value of DECT and mpMRI after the neoadjuvant treatment for pathologic response | 4 years
  Pathological tumour regression grading (Mandard criterion): from 1 to 5 grading.
Disease free survival (DFS) | 4 years
  Survival analysis: Radiologic data predicting DFS.
Overall survival (OS) | 5 years
  Survival analysis: Radiologic data predicting OS.
Likert scales 1-5 | 6 months
  Qualitative image analysis of mpMRI in a supine and prone position
The signal-to-noise Ratio (SNR) | 6 months
  Quantitative image analysis of mpMRI in a supine and prone position.
Contrast-to-noise Ratio (CNR) | 6 months
  Quantitative image analysis of mpMRI in a supine and prone position.

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Dong Zhang, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhen Y, Xie Q, Liu L. Diagnostic Value of Spiral CT and Magnetic Resonance Imaging Scanning in Gastric Cancer and Precancerous Lesions. Scanning. 2022 May 23;2022:3627385. doi: 10.1155/2022/3627385. eCollection 2022. PMID 35795615
- [Background] Giganti F, Orsenigo E, Arcidiacono PG, Nicoletti R, Albarello L, Ambrosi A, Salerno A, Esposito A, Petrone MC, Chiari D, Staudacher C, Del Maschio A, De Cobelli F. Preoperative locoregional staging of gastric cancer: is there a place for magnetic resonance imaging? Prospective comparison with EUS and multidetector computed tomography. Gastric Cancer. 2016 Jan;19(1):216-25. doi: 10.1007/s10120-015-0468-1. Epub 2015 Jan 23. PMID 25614468
- [Background] Borggreve AS, Goense L, Brenkman HJF, Mook S, Meijer GJ, Wessels FJ, Verheij M, Jansen EPM, van Hillegersberg R, van Rossum PSN, Ruurda JP. Imaging strategies in the management of gastric cancer: current role and future potential of MRI. Br J Radiol. 2019 May;92(1097):20181044. doi: 10.1259/bjr.20181044. Epub 2019 Mar 5. PMID 30789792